CLINICAL TRIAL: NCT00375986
Title: A Comparison of Manual vs. Spontaneous Removal of the Placenta at Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 00014248
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Pregnancy; Cesarean Section
Keywords: Cesarean delivery; Placental removal; Blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Manual placental removal at Cesarean delivery
Procedure: Spontaneous placental removal at Cesarean delivery

SUMMARY:
The purpose of this study is to determine if there are differences in operative blood loss with manual vs. spontaneous removal of the placenta during cesarean section.

DETAILED DESCRIPTION:
Patients undergoing scheduled cesarean deliveries are randomized to manual or spontaneous placental removal.

ELIGIBILITY:
Inclusion Criteria:

* All term pregnant women 18 years of age and older undergoing scheduled cesarean delivery at Strong Memorial Hospital.

Exclusion Criteria:

* Prematurity (<37 weeks)
* Preoperative chorioamnionitis
* Vaginal delivery of fetus
* Emergency Cesarean Delivery
* Patient's OB not agreeable to participating in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hematocrit levels (preoperatively and within 48 hours postoperatively)

SECONDARY OUTCOMES:
Number of units of blood transfused intraoperatively and postoperatively
Development of uterine infection (endometritis)
Length of postoperative hospital stay
Operative time

CONTACTS AND LOCATIONS:
Overall Officials: Eva K. Pressman, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States